CLINICAL TRIAL: NCT05325671
Title: Efficacy of Postoperative Pain Control Between Transarticular VS Periartiucular Multimodal Drug Infiltration in Total Hip Arthroplasty: Double-blinded Randomized Control Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 65016
Record Dates: First submitted 2022-04-05; First posted 2022-04-13 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2022-04

CONDITIONS: Pain, Post Operative; Arthroplasty Complications
Keywords: total hip arthroplasty; transarticular multimodal drug infiltration; periarticular multimodal drug infiltration
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transarticular multimodal drug infiltration (Experimental): infiltration the mixture into intraarticular by catheter guided approach
  Interventions: Procedure: transarticular multimodal drug infiltration
- periarticular multimodal drug infiltration (Active Comparator): 3 location of infiltration
  1. hip capsule
  2. gluteus medius and short external rotator
  3. gluteus maximus
  Interventions: Procedure: transarticular multimodal drug infiltration

INTERVENTIONS:
Procedure: transarticular multimodal drug infiltration — as described previously

SUMMARY:
This research aim to improve postoperative outcome in total hip arthroplasty(THA) by using local mixture infiltration as bupivacaine + NSAID + epinephrine + tranxemic acid. In the present time these mixture components has shown to improve THA outcome by aspect of postoperative pain control, postoperative opioid consumption, postoperative bleeding, LOS and postoperative rehabilitation without increasing complication but the accuracy of infiltration technique which gives the best outcome has not been yet discovered.Recently study by Hashimoto et al has risen that these technique can be administrated by both periarticular and intra-articular approach.By considering the complexity of human anatomy around the hip tissue we assume that the intra-articular(transarticular) may given equivalence (may be better) outcome with lowering procedural related complication comparing to periarticular infiltration approach.

ELIGIBILITY:
Inclusion Criteria:

* patient who would go on cemented and cementless THA
* age 45-60 years of age
* voluntary decision exclusion criteria
* bilateral THA
* revision surgery
* history of pelvic and hip surgery previously
* allergy to medication in protocol
* CKD stage 4-5, chronic liver disease with Child Pugh B or C
* pregnancy
* history of hip injection
* U/D
* hypercoagulable state
* abnormal laboratory coagulation study as INR > 1.4 or aPTT > 1.4
* abnormal platelet function
* thrombocytopenia
* PE , DVT, ischemic stroke, CAD/ischemic heart disease
* use of anticoagulant or hormonal usage
* anesthesia by general anesthesia or additional nerve block
* can not understand PCA usage
* use postopertive wound drainage

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale at rest on postoperative day1st and 2nd | 1 week

SECONDARY OUTCOMES:
total morphine consumption in first 24 hours postoperative period via PCA pump | 1 week
total morphine consumption in whole postoperative period | 1 week
length of stay | 1 week
postoperative complication | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Peerapon Nantapong, MD, Study Director — Department of Medical Services Ministry of Public Health of Thailand; Thakrit Chompoosang, MD, Study Chair — Department of Medical Services Ministry of Public Health of Thailand
Locations (1):
- Rajavithi Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Varacallo MA, Luo TD, Johanson NA. Total Hip Arthroplasty Techniques. 2023 Aug 4. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK507864/ PMID 29939641
- [Result] Gaffney CJ, Pelt CE, Gililland JM, Peters CL. Perioperative Pain Management in Hip and Knee Arthroplasty. Orthop Clin North Am. 2017 Oct;48(4):407-419. doi: 10.1016/j.ocl.2017.05.001. Epub 2017 Jun 29. PMID 28870302
- [Result] Chou R, Gordon DB, de Leon-Casasola OA, Rosenberg JM, Bickler S, Brennan T, Carter T, Cassidy CL, Chittenden EH, Degenhardt E, Griffith S, Manworren R, McCarberg B, Montgomery R, Murphy J, Perkal MF, Suresh S, Sluka K, Strassels S, Thirlby R, Viscusi E, Walco GA, Warner L, Weisman SJ, Wu CL. Management of Postoperative Pain: A Clinical Practice Guideline From the American Pain Society, the American Society of Regional Anesthesia and Pain Medicine, and the American Society of Anesthesiologists' Committee on Regional Anesthesia, Executive Committee, and Administrative Council. J Pain. 2016 Feb;17(2):131-57. doi: 10.1016/j.jpain.2015.12.008. PMID 26827847
- [Result] Andersen KV, Pfeiffer-Jensen M, Haraldsted V, Soballe K. Reduced hospital stay and narcotic consumption, and improved mobilization with local and intraarticular infiltration after hip arthroplasty: a randomized clinical trial of an intraarticular technique versus epidural infusion in 80 patients. Acta Orthop. 2007 Apr;78(2):180-6. doi: 10.1080/17453670710013654. PMID 17464604
- [Result] Busch CA, Whitehouse MR, Shore BJ, MacDonald SJ, McCalden RW, Bourne RB. The efficacy of periarticular multimodal drug infiltration in total hip arthroplasty. Clin Orthop Relat Res. 2010 Aug;468(8):2152-9. doi: 10.1007/s11999-009-1198-7. Epub 2009 Dec 18. PMID 20020333
- [Result] Parvataneni HK, Shah VP, Howard H, Cole N, Ranawat AS, Ranawat CS. Controlling pain after total hip and knee arthroplasty using a multimodal protocol with local periarticular injections: a prospective randomized study. J Arthroplasty. 2007 Sep;22(6 Suppl 2):33-8. doi: 10.1016/j.arth.2007.03.034. Epub 2007 Jul 26. PMID 17823012
- [Result] Kurosaka K, Tsukada S, Ogawa H, Nishino M, Nakayama T, Yoshiya S, Hirasawa N. Addition of corticosteroid to periarticular injections reduces postoperative pain following total hip arthroplasty under general anaesthesia: a double-blind randomized controlled trial. Bone Joint J. 2020 Oct;102-B(10):1297-1302. doi: 10.1302/0301-620X.102B10.BJJ-2020-0428.R1. PMID 32993338
- [Result] Tsinaslanidis G, Tsinaslanidis P, Mahajan RH. Perioperative Pain Management in Patients Undergoing Total Hip Arthroplasty: Where Do We Currently Stand? Cureus. 2020 Jul 7;12(7):e9049. doi: 10.7759/cureus.9049. PMID 32782868
- [Result] Becker DE, Reed KL. Local anesthetics: review of pharmacological considerations. Anesth Prog. 2012 Summer;59(2):90-101; quiz 102-3. doi: 10.2344/0003-3006-59.2.90. PMID 22822998
- [Result] El-Boghdadly K, Pawa A, Chin KJ. Local anesthetic systemic toxicity: current perspectives. Local Reg Anesth. 2018 Aug 8;11:35-44. doi: 10.2147/LRA.S154512. eCollection 2018. PMID 30122981
- [Result] Fillingham YA, Ramkumar DB, Jevsevar DS, Yates AJ, Bini SA, Clarke HD, Schemitsch E, Johnson RL, Memtsoudis SG, Sayeed SA, Sah AP, Della Valle CJ. Tranexamic Acid Use in Total Joint Arthroplasty: The Clinical Practice Guidelines Endorsed by the American Association of Hip and Knee Surgeons, American Society of Regional Anesthesia and Pain Medicine, American Academy of Orthopaedic Surgeons, Hip Society, and Knee Society. J Arthroplasty. 2018 Oct;33(10):3065-3069. doi: 10.1016/j.arth.2018.08.002. Epub 2018 Aug 7. No abstract available. PMID 30146350
- [Result] Stoicea N, Moran K, Mahmoud AR, Glassman A, Ellis T, Ryan J, Granger J, Joseph N, Salon N, Ackermann W, Rogers B, Niermeyer W, Bergese SD. Tranexamic acid use during total hip arthroplasty: A single center retrospective analysis. Medicine (Baltimore). 2018 May;97(21):e10720. doi: 10.1097/MD.0000000000010720. PMID 29794747
- [Result] Sukeik M, Alshryda S, Haddad FS, Mason JM. Systematic review and meta-analysis of the use of tranexamic acid in total hip replacement. J Bone Joint Surg Br. 2011 Jan;93(1):39-46. doi: 10.1302/0301-620X.93B1.24984. PMID 21196541
- [Result] Qiu J, Sun X, Zhang W, Ke X, Yang G, Zhang L. Effect of topical tranexamic acid in total hip arthroplasty patients who receive continuous aspirin for prevention of cardiovascular or cerebrovascular events: A prospective randomized study. Orthop Traumatol Surg Res. 2019 Nov;105(7):1327-1332. doi: 10.1016/j.otsr.2019.06.018. Epub 2019 Sep 27. PMID 31570210
- [Result] Ma HH, Chou TA, Tsai SW, Chen CF, Wu PK, Chen WM. The efficacy of intraoperative periarticular injection in Total hip arthroplasty: a systematic review and meta-analysis. BMC Musculoskelet Disord. 2019 Jun 1;20(1):269. doi: 10.1186/s12891-019-2628-7. PMID 31153361
- [Result] Wang Y, Gao F, Sun W, Wang B, Guo W, Li Z. The efficacy of periarticular drug infiltration for postoperative pain after total hip arthroplasty: A systematic review and meta-analysis. Medicine (Baltimore). 2017 Mar;96(12):e6401. doi: 10.1097/MD.0000000000006401. PMID 28328836
- [Result] Hashimoto A, Sonohata M, Kawaguchi A, Kii S, Hirata H, Mawatari M. Comparison of the Effect of Different Local Analgesia Administration Techniques in Total Hip Arthroplasty: A Retrospective Comparative Cohort Study. Pain Res Manag. 2021 Jul 24;2021:9914590. doi: 10.1155/2021/9914590. eCollection 2021. PMID 34349850
- [Result] Nadler SB, Hidalgo JH, Bloch T. Prediction of blood volume in normal human adults. Surgery. 1962 Feb;51(2):224-32. No abstract available. PMID 21936146
- [Result] Tammachote N, Raphiphan R, Kanitnate S. High-dose (3 g) topical tranexamic acid has higher potency in reducing blood loss after total knee arthroplasty compared with low dose (500 mg): a double-blind randomized controlled trial. Eur J Orthop Surg Traumatol. 2019 Dec;29(8):1729-1735. doi: 10.1007/s00590-019-02515-2. Epub 2019 Jul 29. PMID 31359178
- [Result] Gao FQ, Li ZJ, Zhang K, Sun W, Zhang H. Four Methods for Calculating Blood-loss after Total Knee Arthroplasty. Chin Med J (Engl). 2015 Nov 5;128(21):2856-60. doi: 10.4103/0366-6999.168041. PMID 26521781